CLINICAL TRIAL: NCT06396169
Title: The Effect of Yoga Exercises and Callisthenic Exercises on the Quality of Life in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KTOKARACA001
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-04

CONDITIONS: Quality of Life; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Exercise Group (Active Comparator): Yoga Exercises
  Interventions: Other: Yoga Exercise
- Calisthenic Exercise Group (Active Comparator): Calisthenic Exercises
  Interventions: Other: Calisthenic Exercise

INTERVENTIONS:
Other: Yoga Exercise — Yoga Exercises
  Arms: Yoga Exercise Group
Other: Calisthenic Exercise — Calisthenic Exercises
  Arms: Calisthenic Exercise Group

SUMMARY:
In this study, healthy individuals will be asked to do yoga exercises or a calisthenic exercise program. The effect of different exercise programs on quality of life will be investigated.

DETAILED DESCRIPTION:
While yoga was a part of the philosophy of life in India, today it has become widespread as a physical and mental practice and has become a preferred approach to protect and improve physical functions, especially in healthy individuals. The word yoga means "union" and "unity". It is a group of practices or disciplines that mainly include physical movements , special breathing techniques and deep concentration. A study on this subject has shown that Yoga training applied to healthy individuals increases muscle strength, muscle endurance and flexibility, and reduces stress levels.

Calisthenic exercises; These are exercises that are performed by creating resistance only with your body weight, without the need for any equipment or gym. Calisthenic exercises are aerobic and dynamic exercises. Calisthenics exercises are a useful and useful exercise method that can be done at a fast pace, at different intensities, and can also be modified. Calisthenic exercises should be rhythmic and performed by counting. A study on this subject has shown that calisthenic exercises improve muscle strength and balance.

In this study, healthy individuals will be asked to do yoga exercises or a calisthenic exercise program. The effect of different exercise programs on quality of life will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. The ages of 18 - 45
2. No communication problems
3. Not having had a surgical operation in the last 6 months

Exclusion Criteria:

1. Individuals with musculoskeletal system problems that prevent them from exercising
2. Individuals who have respiratory problems when their physical activity increases
3. Individuals with a history of chest pain related and unrelated to physical activity
4. Individuals with chronic diseases

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-05-12 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
36-Item Short Form Survey Instrument | The evaluation will be applied at the baseline and after study completion, an average of 2 months.
  The objective measure of the quality of life. The scale total score from 0 (negative health) to 100 (positive health) .

SECONDARY OUTCOMES:
Positive and Negative Affect Schedule (PANAS) | The evaluation will be applied at the baseline and after study completion, an average of 2 months.
  20-item self- report measure to assess positive affect and negative affect. The total score is calculated by finding the sum of the 10 positive items, and then the 10 negative items. Scores range from 10 - 50 for both sets of items. For the total positive score, a higher score indicates more of a positive affect. For the total negative score, a lower score indicates less of a negative affect.

CONTACTS AND LOCATIONS:
Overall Officials: Osman Karaca, Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not sharing other researchers.